CLINICAL TRIAL: NCT02256904
Title: Biomechanical and Radiostereometric Analysis of the GMK Sphere Primary Total Knee Replacement. A Randomized, Double Blind Comparison of Anatomical Versus Mechanical Alignment in Total Knee Replacement.
Brief Title: RSA and Clinical Comparison of Anatomical and Mechanical Alignment in Total Knee Replacement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Pascal André Vendittoli, clinical researcher, MD, MSc, FRCSC, Maisonneuve-Rosemont Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HMR 01
Record Dates: First submitted 2014-09-30; First posted 2014-10-06 (Estimated); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Personal Satisfaction; Genu Varum
Keywords: Alignment; Kinematic; knee; satisfaction; function; survivorship
MeSH Terms: conditions — Personal Satisfaction; Genu Varum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anatomical (Experimental): 67 subjects will be randomized to receive an Anatomical TKA with the My knee instruments and a GMK sphere device.
  Interventions: Procedure: Anatomical TKA
- Mechanical (Active Comparator): 67 subjects will be randomized to receive a Mechanical TKA with the My knee instruments and the GMK sphere device.
  Interventions: Procedure: Mechanical TKA

INTERVENTIONS:
Procedure: Anatomical TKA — Personalized Medacta plastic cutting blocks will be manufactured according to patient Ct-scan.The anatomical cutting blocks will be design to resurface the femoral and tibial bones to restore each patient's pre-arthritic anatomy within specific margins: maximum of 5 degrees valgus/varus tibial or femoral cut and overall lower limb alignment within +/-3 degrees of varus/valgus). GMK sphere TKA will be implanted using the manufactured cutting blocks.
  Arms: Anatomical
Procedure: Mechanical TKA — Personalized Medacta plastic cutting blocks will be manufactured according to patient Ct-scan. In the mechanical group, femoral and tibial cutting blocks will be designed for a 0-degree angle according to the mechanical axis. Femoral rotation will be aligned with the femoral trans-epicondylar axis. Tibial rotation will follow femoral rotation. GMK sphere TKA will be implanted using the manufactured cutting blocks.
  Arms: Mechanical

SUMMARY:
Current practice in orthopedics is to recommend TKA implantation with the femoral and tibial components perpendicular to their mechanical axis. Therefore, current surgical technique does not replicate natural knee anatomy and biomechanics. An alternative alignment method that attempts to replicate the kinematics of the knee is " kinematic alignment ". The principle behind kinematic alignment is placement of the TKA components so that the orthogonal 3-D orientation of the 3 axes that describe normal knee kinematics is restored to that of the prearthritic knee. Theoretical benefits of kinematic alignment include less ligamentous release to balance the knee intra-operatively, more rapid recovery, better range of motion (ROM), less post-operative pain, better knee biomechanics, and improved patient satisfaction. However, a major concern is that there are no mid- or long-term data on implant survivorship (absence of loosening) in TKA based on "anatomical" implantation. The investigators propose to compare the clinical results of TKA implanted with mechanical alignment (standard practice) to kinematic alignment, in a double-blind, randomized trial.

DETAILED DESCRIPTION:
Problem to be addressed Knee osteoarthritis is a degenerative joint disease that is very prevalent in the general population and can cause significant functional impairment. Total knee arthroplasty (TKA) is the definitive treatment of choice, but rarely accomplishes complete restoration of natural knee biomechanics. Various factors may influence post-operative function: pre-operative state of the knee, patient age, implant position, and design. The natural lower limb anatomy presents a femoral joint surface that is slightly valgus according to its mechanical axis (1-5 degrees) and a tibial joint surface that is slightly varus (1-4 degrees). This combination results in an oblique joint line orientation (1-3 degrees) and a mechanical axis passing near the centre of the knee joint (line between the centre of the femoral head and the centre of the ankle). Natural lower limb alignment helps balancing load between the internal and external knee compartments at heel strike. Current practice in orthopedics is to recommend TKA implantation with the femoral and tibial components perpendicular to their mechanical axis (0 degrees). In addition, in order to maintain ligament balance (a rectangular space) in flexion, external rotation of the femoral implant is suggested (2-5 degrees according to posterior femoral condyle surfaces). Therefore, current surgical technique does not replicate natural knee anatomy and biomechanics. An alternative alignment method that attempts to replicate the kinematics of the knee is " kinematic alignment ". The principle behind kinematic alignment is placement of the TKA components so that the orthogonal 3-D orientation of the 3 axes that describe normal knee kinematics is restored to that of the prearthritic knee. Theoretical benefits of kinematic alignment include less ligamentous release to balance the knee intra-operatively, more rapid recovery, better range of motion (ROM), less post-operative pain, better knee biomechanics, and improved patient satisfaction. However, a major concern is that there are no mid- or long-term data on implant survivorship (absence of loosening) in TKA based on "anatomical" implantation. Because the anatomical alignment differs from the classic mechanical alignment, some authors raised concerns regarding mid-term implant stability with the anatomical implantation technique.

We propose to compare the clinical results of TKA implanted with mechanical alignment (standard practice) to kinematic alignment, in a double-blind, randomized trial. To standardize surgical technique and minimize potential bias, both procedures will be undertaken with personalized instruments built by Medacta, based on each patient's CT-scan.

There are 2 primary objectives of this research. First, implant stability with respect to bone will be measured over time by RSA, and long-term survivorship will be estimated. Second, we will determine if anatomical implantation provides clinical advantages, with respect to knee kinematic analysis, functional performance tests and validated self-reported questionnaires on pain, function and stiffness.

Radiostereometric analysis (RSA) RSA, first developed in Lund, Sweden, is a radiographic technique for accurately assessing implant position relative to host bone. RSA is the gold standard for measuring implant stability in the short-term and predicting implant survivorship in the long-term. It has been implemented for several decades and its safety is well documented. RSA is 10 times more accurate than conventional radiography in analyzing implant migration patterns. Patterns of micromigration exhibited by various prostheses and fixation techniques within the first post-operative year has been shown to predict long-term component fixation to bone.

Knee biomechanical evaluation Estimating the therapeutic efficacy of knee TKA is subjective in current clinical practice because methods of functional biomechanics assessment are complex and difficult to apply. It was suggested that gait measurements should be monitored after surgery for patients with knee osteoarthritis (OA) to evaluate treatment outcome and recovery. KneeKGTM (Emovi Inc., Laval, Quebec, Canada), a simple and minimally-invasive method of measuring 3D knee kinematics, has been developed and is now available commercially. In this system, motion sensors are quasi-rigidly attached to the leg with a non-invasive ancillary system, which reduces errors in skin movement in relation to bone. This measurement tool has been validated by satisfactory assessment of its accuracy and the reproducibility of femoro-tibial 3D kinematics during gait.

Principal research questions

* Compare the migration between anatomically- and mechanically-aligned implants at 2 years and predict the long-term survivorship of total knee prostheses inserted with these two techniques.
* Compare the clinical results of anatomical and mechanical total knee alignment with self reported pain, function and stiffness questionnaire scores.
* Compare knee kinematics between the 2 groups and identify biomechanical markers that explain subjective differences (if found with clinical scores).
* Compare kinematics measured with the 2 techniques to those of asymptomatic knees.
* Determine if anatomical alignment offers some technical benefits (reduced intra-operative ligament balance and ligaments releases) compared to a mechanical alignment technique.
* Compare post-operative rehabilitation in both groups (flexion, extension, straight leg raising, walking without assistance, etc.).

Hypothesis TKA implanted with with anatomical alignment will provide better clinical outcomes and knee kinematics closer to normal than TKA implanted with a mechanical alignment technique, Implant longevity will show similar micro migration patterns between the two groups as measured by RSA up to 2 years after implantation thereby predicting that long-term implant survivorship will be similar in both groups.

Why is this trial needed now? Current technological advances in knee arthroplasty surgery have allowed surgeons to implant TKA with considerable accuracy. We however are not sure if the position we are placing the knee in is the "correct" position for most patients. It is thought that the relatively high percentage of patients that are not completely satisfied with the outcome of their knee replacement may have the implants in a suboptimal position for that individual patient. The traditional mechanical alignment may not be the optimal position for these patients. The anatomical alignment technique may reduce the percentage of dissatisfied patients. Implant companies with this technology are currently marketing this to surgeons and patients without clinical data to support this claim. There is also the possibility that placing an artificial knee joint in an anatomic position may impart a negative impact on longevity of the implant, thus increasing early revision rates and the significant health costs associated with this. Thus it becomes mandatory to evaluate this new technology before its widespread adoption in clinical practice to determine the real benefits or disadvantages of changing from a successful clinical practice (mechanical alignment) used over the last 40 years.

Trial results This proposed clinical trial will have a direct impact on patient care if it demonstrates that anatomical alignment TKA provides better clinical results than mechanical alignment TKA and similar migration patterns measured by RSA. Then the use of anatomic alignment may become the gold standard for TKA procedures. Lacking accurate investigation and surgical tools, anatomical alignment was abandoned in the early TKA era. Mechanical alignment was selected to minimize errors and secondary failures. With novel technologies (personalized instruments built on MRI), anatomical alignment might be the best way to replicate knee biomechanics and improve patient outcomes after TKA. The proposed study will allow us to establish the real value of anatomical alignment and its safety.

ELIGIBILITY:
Inclusion Criteria:

1. Patient qualifies for primary TKA
2. Patient understands the study conditions
3. Patient is capable of giving informed consent

Exclusion Criteria:

1. Other joint damage of the lower limbs
2. Extra-articular knee deformation of the lower limb
3. Hip arthroplasty on the surgical side
4. Contraindication to CT-scan
5. Acute or chronic infection of the lower limb
6. Progressive local or systemic infection
7. Alcohol or drug abuse
8. Psychiatric illness/mental disorder
9. Pregnancy
10. Less than 18 years of age
11. Known allergy to the implant materials
12. Muscular loss, neuromuscular disease or vascular deficiency of the affected limb making the operation unjustifiable
13. Any neuromuscular disorder
14. Severe instability secondary to advanced destruction of osteochondral structures or loss of integrity of the lateral ligament

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2015-04-13 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Component migration measured with Radiostereophotometry | 2 years
  In the first 40 cases (20 in each group), we will compare the migration with a RSA system between anatomically- and mechanically-aligned implants at 2 years and predict the long-term survivorship of total knee prostheses inserted with these two techniques.

SECONDARY OUTCOMES:
Clinical scores | 2 years
  In all randomized subject, we will compare the clinical results of anatomical and mechanical total knee alignment with self reported pain, function and stiffness questionnaire scores. Validated clinical scores will be used: WOMAC, KOOS and SF-12
Knee kinematics measured with the Knee KG (Emovi inc.) | 2 years
  In all randomized cases, we will compare post operative knee kinematics with the Knee KG system (Emovi inc) between the 2 groups and identify biomechanical markers that explain subjective differences (if found with clinical scores).
Technical benefits | 1 month
  In all randomized cases, we will determine if anatomical alignment offers some technical benefits (reduced intra-operative ligament balance and ligaments releases) compared to a mechanical alignment technique.
Rehabilitation | 1 month
  In all cases, we will compare post-operative rehabilitation in both groups (flexion, extension, straight leg raising, walking without assistance, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Andre Vendittoli, MD, MSc, Principal Investigator — Research Director and surgeon
Locations (1):
- Hopital Maisonneuve Rosemont, Montreal, Quebec, Canada